CLINICAL TRIAL: NCT06720467
Title: Role of Immunotherapy in the Treatment of Eyelid Viral Papilloma
Brief Title: Immunotherapy in Eyelid Viral Papilloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Marwa Ahmed Khairy Elsayed Essa, Principle investigator, lecturer of ophthalmology, Faculty of Medicine, Zagazig University, Zagazig, Egypt, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: immunotherapy in eyelid warts
Record Dates: First submitted 2024-12-01; First posted 2024-12-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-12

CONDITIONS: Eye Infections
Keywords: eyelid warts, candida antigen, eyelid papilloma
MeSH Terms: conditions — Eye Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- patients with eyelid warts will receive treatment in the form of intralesional injection of Candida (Experimental): Intralesional injection of 0.2 ml of 1/1000 solution of Candida albicans antigen using an insulin syringe directly into the warts; Candida albicans 1:20 w/v 10 ml vial (Allergy Laboratories, INC. Oklahoma City, USA.). The same injection was repeated every 2 weeks until complete clearance for a maximum of six treatment sessions.
  Interventions: Biological: Intralesional injection of Candida albicans 1:20 w/v 10 ml vial (Allergy Laboratories, INC. Oklahoma City, USA.)

INTERVENTIONS:
Biological: Intralesional injection of Candida albicans 1:20 w/v 10 ml vial (Allergy Laboratories, INC. Oklahoma City, USA.) — Intralesional injection of 0.2 ml of 1/1000 solution of Candida albicans antigen using an insulin syringe directly into the warts; Candida albicans 1:20 w/v 10 ml vial (Allergy Laboratories, INC. Oklahoma City, USA.). The same injection was repeated every 2 weeks until complete clearance for a maximum of six treatment sessions.

SUMMARY:
intralesional injection of Candida antigens for treating eyelid warts is supposed to have less destructive effect than other surgical interventions

DETAILED DESCRIPTION:
Despite many surgical and interventional modalities of treating ocular warts, all have a destructive nature for this delicate tissue with a high recurrence rate. intralesional injection of Candida antigens was suggested to be an effective and safe treatment for such a condition aim: Providing safe and effective treatment of ocular wart. objective:

1. To determine the efficacy of intralesional injection of Candida antigens in the treatment of eyelids wart
2. To determine the safety of intralesional injection of Candida antigens in the treatment of eyelids wart
3. To report complications of intralesional injection of Candida antigens in the treatment of eyelids wart

ELIGIBILITY:
Inclusion Criteria:

* patients with cutaneous eyelid viral warts whether single or multiple, with no concurrent systemic or topical treatment for warts. Patients aged more than 12 years, with sensitivity test, showed induration less than or equal to five mm. and patients can understand and comply with the requirements of the trials.

Exclusion Criteria:

* pregnancy, breastfeeding, patients with immunodeficiency; like diabetics. In addition, patients with a history of hypersensitivity to any used component in this trial, asthma, or allergic skin diseases. Moreover, patients on any treatment modality for warts at least 1 month before the start of the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-11 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
complete response | after maximum 6 treatment sessions of intralesional injection with 2 weeks between the successive sessions
  to report the complete response defined by the efficacy of intralesional injection of Candida antigen in achieving complete disappearance of eyelid warts and return to normal skin

SECONDARY OUTCOMES:
partial response | after maximum 6 treatment sessions of intralesional injection with 2 weeks between the successive sessions
  to report Partial response which will be considered when wart regress in size by 50%-99%.
Failure | after maximum 6 treatment sessions of intralesional injection with 2 weeks between the successive sessions
  to report failure which will be considered if less than 50% decrease in wart size.
complications | after maximum 6 treatment sessions of intralesional injection with 2 weeks between the successive sessions
  to report any complications in the form of hypersensitivity reaction, erythema, or induration

CONTACTS AND LOCATIONS:
Overall Officials: Ayman Marie, Professor, Principal Investigator — Professor of Medical Microbiology and Immunology, Faculty of Medicine, Zagazig University, Egypt; Ghada Boghdadi, Professor, Study Chair — Professor of Medical Microbiology and Immunology, Faculty of Medicine, Zagazig University, Egypt
Locations (1):
- Zagazig University, Zagazig, Zagazig, Egypt

REFERENCES:
- [Background] Marei A, Nofal A, Alakad R, Abdel-Hady A. Combined bivalent human papillomavirus vaccine and Candida antigen versus Candida antigen alone in the treatment of recalcitrant warts. J Cosmet Dermatol. 2020 Mar;19(3):758-762. doi: 10.1111/jocd.13077. Epub 2019 Jul 22. PMID 31328869
- [Background] Aldahan AS, Mlacker S, Shah VV, Kamath P, Alsaidan M, Samarkandy S, Nouri K. Efficacy of intralesional immunotherapy for the treatment of warts: A review of the literature. Dermatol Ther. 2016 May;29(3):197-207. doi: 10.1111/dth.12352. Epub 2016 Mar 15. PMID 26991521
- [Background] Shaker ESE, Doghim NN, Hassan AM, Musafa SS, Fawzy MM. Immunotherapy in cutaneous warts: comparative clinical Study between MMR vaccine, tuberculin, and BCG Vaccine. J Cosmet Dermatol. 2021 Aug;20(8):2657-2666. doi: 10.1111/jocd.13921. Epub 2021 Jan 6. PMID 33410249